CLINICAL TRIAL: NCT01514305
Title: Observational Study to Evaluate the Effectiveness and Safety Study of the Dexcom G4™ Continuous Glucose Monitoring System
Status: Completed | Type: Observational
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTL900830
Record Dates: First submitted 2011-11-28; First posted 2012-01-23 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type 1 Diabetes Mellitus (TIDM)Type 2 Diabetes Mellitus (T2DM): Adults that have been diagnosed with insulin-requiring diabetes and are on multiple daily injections (MDI) or Continuous Subcutaneous Insulin Infusion (CSII) insulin therapy;

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of the Dexcom G4 System when used as an adjuvant to blood glucose testing.

Device performance will be primarily evaluated in terms of the proportion of glucose values within a pre-specified range compared to reference values.

Safety data of the G4 System will also be collected vis-a-vis adverse event reporting characterized by the incidence and severity of Serious Adverse Device Events, and Adverse Device Events experienced by study participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Have been diagnosed with insulin-requiring diabetes
3. Abstain from injecting insulin or wear an insulin pump insertion set within 3 inches from the sensor site during sensor wear;
4. Insert sensors on their own and wear 2 systems simultaneously;
5. Use only the blood glucose meter provided for all blood glucose measurements performed during sensor wear and not allow others to use this meter during the study;
6. Participate in one in-clinic session comprising of fingersticks per hour and have blood draws for the entire in-clinic session;
7. Have an intravenous catheter inserted for 4 blood draws per hour
8. Willing to perform SMBG during home use with the meter provided;
9. Refrain from the use of acetaminophen during sensor wear period and the day prior to sensor insertion;
10. Speak, read, and write English;
11. Willing and able to be compliant with provisions laid out in this protocol.

Exclusion Criteria:

1. Have extensive skin changes/diseases that preclude wearing devices on normal skin (e.g., extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis) at the proposed wear sites;
2. Allergy to medical-grade adhesives;
3. Pregnant as demonstrated by a positive pregnancy test within 72 hours of sensor insertion,
4. Dialysis treatment;
5. Hematocrit that is outside the range of 30-55% at screening visit;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects that fit the inclusion criteria will be chosen from the general population
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Absolute Relative Difference (%) to Reference Standard | one time measure (day 1)
  The primary objective is to characterize the System performance with respect to laboratory reference venous sample measurements. The device performance will be primarily evaluated in terms of point and rate accuracy of the G4 System in reference to YSI. The point accuracy is measured as the proportion of G4 System values that are within ±20% of YSI reference value for glucose levels >80 mg/dL and ±20 mg/dL at YSI glucose levels <80 mg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: David Price, MD, Study Director — DexCom, Inc.
Locations (1):
- Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho, United States